CLINICAL TRIAL: NCT06332781
Title: Intravesical Gentamicin to Prevent Recurrent UTI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2126175 // CTR grant U54GM1156
Record Dates: First submitted 2023-12-13; First posted 2024-03-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Uti
MeSH Terms: conditions — Urinary Tract Infections | interventions — Gentamicins; Nitrofurantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care
  Interventions: Drug: Nitrofurantoin
- Experimental (Experimental): Gentamicin
  Interventions: Drug: Gentamicin

INTERVENTIONS:
Drug: Gentamicin — administered via bladder
  Arms: Experimental
Drug: Nitrofurantoin — administered PO
  Arms: Standard of Care

SUMMARY:
Feasibility assessment of intravesical gentamicin instillation (putting antibiotics directly into the bladder) versus the current standard of care of oral nitrofurantoin prophylaxis (taking a low dose of antibiotics by mouth every day) to prevent recurrent urinary tract infections (UTI)

DETAILED DESCRIPTION:
The overall goal of this project is to assess the feasibility of a larger trial investigating the use of intravesical gentamicin instillation (putting antibiotics directly into the bladder) versus the current standard of care of oral nitrofurantoin prophylaxis (taking a low dose of antibiotics by mouth every day). Investigators plan to gain patient perspective regarding preferences for study design and assess associations between the treatments with changes in the postmenopausal urinary microbiome (urobiome).

ELIGIBILITY:
Inclusion criteria:

* Postmenopausal
* 2 UTIs in 6 months
* desire to start antibiotic prophylaxis to prevent UTIs

Exclusion criteria:

* Parkinsons disease
* myasthenia gravis
* renal failure
* liver failure
* bladder pain syndrome
* multiple negative urine cultures associated with UTI symptoms (>/= 3)
* bladder Botox treatments in the past
* treatment planned for UI and prolapse
* unevaluated microscopic hematuria
* history of kidney stones
* no antibiotics within 4 weeks
* most recent weight <40kg (88.18lbs)
* surgically altered urinary tract (urinary diversion, phalloplasty, etc)
* allergy or hypersensitivity to either of the study medications or medications in the same family including but not limited to: amikacin, kanamycin, neomycin, paromomycin, streptomycin, tobramycin.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Enrollment: 30 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Assess feasibility of trial recruitment | 3 months
  measure screening ratio (number of people screened versus number enrolled)
Examine treatment compliance | 3 months
  compare medication compliance between groups, as measured by weekly self-reported number of doses taken in the oral medication group and attendance at installation visits in the intravesical gentamicin group
Examine trial retention | 3 months
  compare the proportion of participants retained in each group

SECONDARY OUTCOMES:
culture-proven UTIs | 3 months
Patient reported outcome measures | 6 weeks, 3 months
  UTI Symptom Assessment
Patient reported outcome measures | 6 weeks, 3 months
  recurrent UTI symptom scale
Patient reported outcome measures | 6 weeks, 3 months
  recurrent UTI impact questionaire
Patient reported outcome measures | 6 weeks, 3 months
  short-form-36
Patient reported outcome measures | 6 weeks, 3 months
  general anxiety disorder-7
Patient reported outcome measures | 6 weeks, 3 months
  patient health questionnaire

OTHER OUTCOMES:
urobiome analysis | 6 weeks, 3 months
  bacterial presence
urobiome analysis | 6 weeks, 3 months
  antimicrobial resistance gene presence

CONTACTS AND LOCATIONS:
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No